CLINICAL TRIAL: NCT00331045
Title: Clinical Evaluation of Alvimopan (SB767905) on Constipation and Related Symptoms Associated With Opioid -A Placebo-controlled Double-blind Study in Cancer Patients-
Brief Title: Clinical Evaluation Of Alvimopan (SB767905) On Constipation And Related Symptoms Associated With Opioid
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Subject registration did not proceed as expected; difficult to complete within scheduled time frame; prematurely terminated w/ 21 subjects randomized.
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABD102965
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2009-09

CONDITIONS: Cancer; Constipation
Keywords: Opioids; cancer; constipation
MeSH Terms: conditions — Neoplasms; Constipation | interventions — alvimopan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Alvimopan 0.25 mg/yday (Experimental)
  Interventions: Drug: alvimopan
- Alviompan 0.5 mg/day (Experimental)
  Interventions: Drug: Alvimopan 0.5 mg/day
- Alvimopan 1 mg/day (Experimental)
  Interventions: Drug: Alvimopan 1 mg/day

INTERVENTIONS:
Drug: alvimopan — 0.25 mg/day
  Other Names: SB767905
  Arms: Alvimopan 0.25 mg/yday
Drug: Placebo
  Arms: Placebo
Drug: Alvimopan 0.5 mg/day
  Arms: Alviompan 0.5 mg/day
Drug: Alvimopan 1 mg/day
  Arms: Alvimopan 1 mg/day

SUMMARY:
This study is intended to investigate the recommended dose of alvimopan in doses 0.25mg/day (0.25mg, OD), 0.5mg/day (0.25mg, BID) or 1mg/day (0.5mg, BID) or placebo for 3 weeks in patients who receive opioids for the management of cancer pain and develop constipation, by giving overall consideration to the efficacy and safety data in each treatment group. Also, efficacy and safety data of alvimopan in the recommended dose group will be compared with those of placebo and to confirm alvimopan's safety and efficacy.

ELIGIBILITY:
Inclusion criteria:

* Have cancer.
* Taking opioid therapy for continued intractable pain.
* Experiencing less bowel movement frequency compared to that before the opioid treatment.
* Must meet the protocol-definition of opioid-induced constipation.

Exclusion criteria:

* Gastrointestinal or pelvic disorders known to affect gastrointestinal functions or induce bowel transit disorder and ileus.
* Subjects, who in the investigator's opinion, have gastrointestinal dysfunction predominantly due to causes other than the use of opioids.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-04; Primary Completion 2006-10 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline during the 1-week Pre-Treatment Period in average weekly bowel movement with no rescue laxative use in the previous 24 hours Frequency during the 3-week Treatment Period

SECONDARY OUTCOMES:
Proportion of responders for OBD global improvement Changes in weekly subjective bowel movement symptoms Changes in weekly constipation symptoms questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline